CLINICAL TRIAL: NCT00481520
Title: A Randomized, Double-blind, Placebo-controlled, Safety, Tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD) Trial of Multiple Ascending Fixed Doses of SAM-531 in Subjects With Mild to Moderate Alzheimer's Disease.
Brief Title: Study Evaluating the Safety,Tolerability, PK and PD of SAM-531 in the Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 3193A1-2000
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2008-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: SAM-531
- 2 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: SAM-531
  Arms: 1
Other: placebo
  Arms: 2

SUMMARY:
The primary purpose of the study is to assess whether SAM-531, an investigational drug, is safe and well tolerated, compared with placebo (a medically inactive substance), in subjects with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria

1. Signed and dated written informed consent obtained from the subject or the subject's legally authorized representative (LAR) or next of kin (if applicable), in accordance with the local regulations. The subject's caregiver must also consent to participate in the study.
2. Diagnosis of probable Alzheimer's Disease according to National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
3. Men and postmenopausal or surgically sterile women aged from 50 to 90 inclusive. Postmenopausal women must have had 12 months of spontaneous amenorrhea. Surgically sterile women are defined as having a hysterectomy, bilateral ovariectomy [oophorectomy], or bilateral tubal ligation. Men who are sexually active will need to agree to use a form of contraception that is satisfactory as per the investigator.
4. Able to participate in all scheduled evaluations with a high probability of completing all required procedures and neuropsychological tests.

Exclusion Criteria

1. Significant neurological disease other than Alzheimer's disease, which may affect cognition (eg, epilepsy, Parkinson disease).
2. Current diagnosis of a major depressive disorder or other major psychiatric symptom according to the criteria of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Version (DSM-IV-TR).
3. Current clinically significant systemic illness, which is likely to deteriorate or affect the subject's safety, influence cognitive assessment or ability to complete the study.
4. Any clinically important deviation from normal limits in physical and neurological examination, vital signs, on electrocardiogram (ECG) or clinical laboratory test results that could compromise the study or be detrimental to the subject.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Routine safety and tolerability will be evaluated. | 28 days

SECONDARY OUTCOMES:
This study will also investigate the pharmacokinetics(PK, how the drug is metabolized) and pharmacodynamics (PD, how the drug affects bodily and mental function) of SAM-531 compared to placebo. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (7):
- United States (7):
  - Delray Beach, Florida
  - Hallandale, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Long Branch, New Jersey
  - New York, New York
  - Bennington, Vermont